CLINICAL TRIAL: NCT05064189
Title: Protection of Corneal Epithelium Using Chitosan-N-acetylcysteine Eye Drops During and/or After Cataract Surgery: a Pilot Study
Brief Title: Protection of Corneal Epithelium Using Chitosan-N-acetylcysteine Eye Drops During and/or After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lacrimera Staining
Record Dates: First submitted 2021-08-31; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): 15 patients will be included in group 1 (no additional treatment)
- Group 2 (Experimental): 15 patients will be in group 2 (treatment directly after cataract surgery in the surgical theatre)
  Interventions: Device: Lacrimera
- Group 3 (Experimental): 15 patients will receive treatment after local anaesthesia (pre-operatively) and directly after cataract surgery (group 3)
  Interventions: Device: Lacrimera

INTERVENTIONS:
Device: Lacrimera — A new preservative-free formulation of eye drops consists of a novel biopolymer, chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria), which electrostatically binds to the mucine layer of the tear film forming a glycocalyx-like structure.
  Arms: Group 2; Group 3

SUMMARY:
The aim of this study is to assess if treatment with Lacrimera® eye drops (Croma-Pharma GbmH, Leobendorf, Austria) during and/ or after cataract surgery has a positive effect on the ocular surface compared to control group.

DETAILED DESCRIPTION:
Prior to surgery, pre-assessment measurements will be performed in the same fashion as for non-study patients. Patients will be randomized to one of the 3 groups in a 1:1:1 fashion using an online randomization tool (www.randomizer.org, list randomizer).

Surgery is performed in topical anaesthesia. Right after topical anaesthesia, patients allocated to Group 3 will receive 1 drop of Lacrimera® in the study eye. Injection of viscoelastic substance (OVD), capsulorhexis, phacoemulsification, and coaxial irrigation/ aspiration of cortical material are performed as standard procedure. After IOL implantation the OVD will be removed and at the end of the surgery, stromal hydration will be performed to the incision as a routine procedure to seal the wound. Right after the wound is sealed, patients allocated to group 2 and group 3 will receive 1 drop of Lacrimera® in the study eye. Postoperative standard medication (Bromfenac gtt., twice a day for 4 weeks) will be prescribed for all groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 or older
* Scheduled for cataract surgery
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX), Intraoperative Floppy Iris Syndrome (IFIS), cornea pathology (e.g. corneal scars, etc.)
* Usage of eye drops other than lubricants (e.g. antibiotics, steroids, cyclosporin-A)
* Previous ocular surgery or trauma in the study eye within 6 months of the cataract surgery
* Active ocular infection or inflammation
* Pregnancy (pregnancy test will be taken in women of reproductive age)
* Subjects with surgery longer than 30 minutes will be excluded and replaced

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Difference in National Eye Institute Grading Scale (NEI Score) | Day 0
  Difference in National Eye Institute Grading Scale (NEI Score) between baseline and 1 hour post cataract surgery

SECONDARY OUTCOMES:
Difference in NEI Score between all visits post-operatively in the different groups | 7 days +/- 1 day
  Difference in NEI Score between all visits post-operatively in the different groups
Difference in break-up time and non-invasive break-up time between the groups at all visits | 7 days +/- 1 day
  Difference in break-up time and non-invasive break-up time between the groups at all visits
Difference in NEI Score between the groups at all visits | 7 days +/- 1 day
  Difference in NEI Score between the groups at all visits
Subjective complaints using OSDI score | 7 days +/- 1 day
  Subjective complaints in the 3 groups using OSDI score
Difference in break-up time and non-invasive break-up time between baseline and 1 week post-operatively in the different groups | 7 days +/- 1 day
  Difference in break-up time and non-invasive break-up time between baseline and 1 week post-operatively in the different groups
Difference in number of MMP-9 positive eyes | 7 days +/- 1 day
  Difference in number of MMP-9 positive eyes before surgery and 1 week after surgery in the different groups
Subjective complaints using VAS | 7 days +/- 1 day
  Subjective complaints in the 3 groups using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, PrimUnivPrDr, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No